CLINICAL TRIAL: NCT01760993
Title: A Phase 3, Long-term, Open-label, Multicenter, 52-week, Flexible-dose Safety Study of SPD489 as Adjunctive Treatment to Established Maintenance Doses of Antipsychotic Medications on Negative Symptoms in Clinically Stable Adults Who Have Persistent Predominant Negative Symptoms of Schizophrenia
Brief Title: Long-term Safety of SPD489 When Added to Stable Doses of Antipsychotic Medications in Clinically Stable Adults With Negative Symptoms of Schizophrenia
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study was discontinued due to non-safety related business prioritization decisions. No subjects were randomized.
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SPD489-336; 2012-003920-18 (EudraCT Number)
Record Dates: First submitted 2013-01-02; First posted 2013-01-04 (Estimated); Results first posted 2014-05-29 (Estimated); Last update posted 2021-06-22 (Actual); Status verified 2021-05

CONDITIONS: Schizophrenia
Keywords: Not Required
MeSH Terms: conditions — Schizophrenia | interventions — Lisdexamfetamine Dimesylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- SPD489 (Experimental)
  Interventions: Drug: SPD489

INTERVENTIONS:
Drug: SPD489 — Once-daily oral optimized doses of SPD489 (either 40 mg, 80 mg, 100 mg, 120 mg, 140 mg, or 160 mg) for 52 weeks
  Other Names: lisdexamfetamine dimesylate, LDX, Vyvanse

SUMMARY:
The primary purpose of this study is to determine if the long-term use of SPD489 (40, 80, 100, 120, 140, and 160mg) administered as a daily morning is safe and tolerable.

DETAILED DESCRIPTION:
Not required

ELIGIBILITY:
Inclusion Criteria:

* 18 to 65 years of age
* Has a reliable informant (eg, family member, social worker, caseworker, or nurse that spends >4 hours/week with the subject)
* Fixed home/place of residence and can be reached by telephone
* On a stable dose of antipsychotic medications
* Able to swallow capsules

Exclusion Criteria:

* -Taking lithium, carbamazepine, lamotrigine, gabapentin, cholinesterase inhibitors, modafinil, or other stimulants such as methylphenidate and other amphetamine products
* Treated with clozapine in past 30 days
* Lifetime history of stimulant, cocaine, or amphetamine abuse or dependence
* History of seizures (other than infantile febrile seizures), any tic disorder, or current diagnosis and/or a known family history of Tourette's Disorder, serious neurological disease, history of significant head trauma, dementia, cerebrovascular disease, Parkinson's disease, or intracranial lesions
* Uncontrolled hypertension
* History of thyroid disorder that has not been stabilized on thyroid medication
* Glaucoma
* Pregnant or nursing
* Subject has received an investigational product or participated in a clinical study within 30 days

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2013-02-01 (Actual); Primary Completion 2013-04-01 (Actual); Study Completion 2013-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (2):
- United States (2):
  - SP Research PLLC/Oklahoma Clinical Research Center, Oklahoma City, Oklahoma
  - CRI Lifetree, Philadelphia, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Study was discontinued due to non-safety related business prioritization decisions. No subjects were randomized
Period: Overall Study
Arm/Group | SPD489
Started | 0
Completed | 0
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Study was discontinued due to non-safety related business prioritization decisions. No subjects were randomized
Arm/Group | SPD489
Number analyzed (Participants) | 0
Age, Categorical
Sex: Female, Male
Region of Enrollment

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Positive and Negative Syndrome Scale (PANSS) Scores at 52 Weeks
Time Frame: Basline and 52 weeks
Population: Study was discontinued due to non-safety related business prioritization decisions. No subjects were randomized
Arm/Group | SPD489
Number analyzed (Participants) | 0

2. Primary Outcome: Change From Baseline in Cognitive Test Battery (CogState Battery) Score at 52 Weeks
Time Frame: Baseline and 52 weeks
Population: Study was discontinued due to non-safety related business prioritization decisions. No subjects were randomized
Arm/Group | SPD489
Number analyzed (Participants) | 0

3. Primary Outcome: Columbia-Suicide Severity Rating Scale (C-SSRS)
Time Frame: Up to 52 weeks
Population: Study was discontinued due to non-safety related business prioritization decisions. No subjects were randomized
Arm/Group | SPD489
Number analyzed (Participants) | 0

4. Primary Outcome: Change From Baseline in Calgary Depression Scale for Schizophrenia (CDSS) at 52 Weeks
Time Frame: Baseline and 52 weeks
Population: Study was discontinued due to non-safety related business prioritization decisions. No subjects were randomized
Arm/Group | SPD489
Number analyzed (Participants) | 0

5. Primary Outcome: Change From Baseline in Simpson Angus Scale (SAS) Total Score at 52 Weeks
Time Frame: Baseline and 52 weeks
Population: Study was discontinued due to non-safety related business prioritization decisions. No subjects were randomized
Arm/Group | SPD489
Number analyzed (Participants) | 0

6. Primary Outcome: Change From Baseline in Barnes Akathisia Scale (BAS) Total Score at 52 Weeks
Time Frame: Baseline and 52 weeks
Population: Study was discontinued due to non-safety related business prioritization decisions. No subjects were randomized
Arm/Group | SPD489
Number analyzed (Participants) | 0

7. Primary Outcome: Change From Baseline in the Abnormal Involuntary Movement Scale (AIMS) at 52 Weeks
Time Frame: Baseline and 52 weeks
Population: Study was discontinued due to non-safety related business prioritization decisions. No subjects were randomized
Arm/Group | SPD489
Number analyzed (Participants) | 0

8. Primary Outcome: Change From Baseline in Clinical Evaluation of Harmful Behavior (CEHB) Scale at 52 Weeks
Time Frame: Baseline and 52 weeks
Population: Study was discontinued due to non-safety related business prioritization decisions. No subjects were randomized
Arm/Group | SPD489
Number analyzed (Participants) | 0

9. Primary Outcome: Change From Baseline in Amphetamine Cessation Symptom Assessment (ACSA) Total Score at 52 Weeks
Time Frame: Baseline and 52 weeks
Population: Study was discontinued due to non-safety related business prioritization decisions. No subjects were randomized
Arm/Group | SPD489
Number analyzed (Participants) | 0

10. Secondary Outcome: Change From Baseline in Negative Symptom Assessment (NSA-16) Total Score at 52 Weeks
Time Frame: Baseline and 52 weeks
Population: Study was discontinued due to non-safety related business prioritization decisions. No subjects were randomized
Arm/Group | SPD489
Number analyzed (Participants) | 0

11. Secondary Outcome: Change From Baseline in the Personal and Social Performance (PSP) Scale Score at 52 Weeks
Time Frame: Baseline and 52 weeks
Population: Study was discontinued due to non-safety related business prioritization decisions. No subjects were randomized
Arm/Group | SPD489
Number analyzed (Participants) | 0

12. Secondary Outcome: Clinical Global Impression-Schizophrenia Severity of Illness (CGI-SCH-S) Scale
Time Frame: Baseline and week 52
Population: Study was discontinued due to non-safety related business prioritization decisions. No subjects were randomized
Arm/Group | SPD489
Number analyzed (Participants) | 0

13. Secondary Outcome: Clinical Global Impression-Schizophrenia Degree of Change (CGI-SCH-C) Scale
Time Frame: Up to 52 weeks
Population: Study was discontinued due to non-safety related business prioritization decisions. No subjects were randomized
Arm/Group | SPD489
Number analyzed (Participants) | 0

14. Secondary Outcome: Change From Baseline in Social Functioning Scale (SFS) at 52 Weeks
Time Frame: Baseline and 52 weeks
Population: Study was discontinued due to non-safety related business prioritization decisions. No subjects were randomized
Arm/Group | SPD489
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Description: Study was discontinued due to non-safety related business prioritization decisions. No subjects were randomized
Arm/Group | SPD489
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
Study was discontinued due to non-safety related business prioritization decisions. No subjects were randomized

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.